CLINICAL TRIAL: NCT05131581
Title: The First Visit for Gynaecological Screening - How do we Make it as Valuable as Possible?
Brief Title: Strategies to Improve the Experience of Gynaecological Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Sophiahemmet University (Other); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Jenny Stern, PhD, Associate Professor, Uppsala University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UU-RLP-Cellprov-2021
Record Dates: First submitted 2021-11-01; First posted 2021-11-23 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
Keywords: Health promotion; Patient experience; Cervical screening test
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (No Intervention): Standard care for cervical screening test (CST) at the midwifery clinic (control group)
- Group 2 (Experimental): Standard care for CST at the youth clinic (intervention group 1)
  Interventions: Other: Changed clinical context
- Group 3 (Experimental): Standard care for CST at the youth clinic with extra time allotted (intervention group 2)
  Interventions: Other: Changed clinical context; Behavioral: Extra time allotted
- Group 4 (Experimental): Standard care for CST at the youth clinic with extra time allotted and the RLP-information (intervention group 3)
  Interventions: Other: Changed clinical context; Behavioral: Extra time allotted; Behavioral: RLP-information

INTERVENTIONS:
Other: Changed clinical context — Changed clinical context: from midwifery clinic to youth clinic
  Arms: Group 2; Group 3; Group 4
Behavioral: Extra time allotted — Extra time allotted for each visit for CST
  Arms: Group 3; Group 4
Behavioral: RLP-information — Midwife-initiated discussion of the Reproductive Life Plan
  Arms: Group 4

SUMMARY:
The aim is to evaluate different strategies to improve the experience and effect of the first visit for a cervical screening test (CST).

1. How do the context and the allotted time for the first visit for a CST affect women's i) experience of CST ii) knowledge of and attitudes towards CST and cervical cancer and iii) attitude towards contacting a midwife regarding sexual and reproductive health in the future
2. What effects do the RLP have, when used as a starting point for counselling at the first visit for a CST, on women's i) experience of CST ii) knowledge of and attitudes towards CST and cervical cancer iii) attitude towards contacting a midwife regarding sexual and reproductive health in the future and iv) knowledge of and attitudes towards fertility and preconception health

Method: cluster randomised control trial evaluating the effect of different strategies, including RLP-based information, to improve the experience and effect of the first visit for a CST.

DETAILED DESCRIPTION:
The aim is to evaluate different strategies to improve the experience and effect of the first visit for a cervical screening test (CST).

1. How do the context and the allotted time for the first visit for a CST affect women's i) experience of CST ii) knowledge of and attitudes towards CST and cervical cancer and iii) attitude towards contacting a midwife regarding sexual and reproductive health in the future
2. What effects do the RLP have, when used as a starting point for counselling at the first visit for a CST, on women's i) experience of CST ii) knowledge of and attitudes towards CST and cervical cancer iii) attitude towards contacting a midwife regarding sexual and reproductive health in the future and iv) knowledge of and attitudes towards fertility and preconception health

The study is a cluster randomized controlled trial evaluating different strategies, RLP-based information, to improve the experience and effect of the first visit for a cervical screening test (CST). The study will be conducted in a strategically chosen area which includes both rural and urban areas, high and low socioeconomic status and high and low percentage of immigrant visitors. The study is conducted in four steps: 1. Standard care for CST at the midwifery clinic (control group) 2. Standard care for CST at the youth clinic (intervention group 1) 3. Standard care for CST at the youth clinic with extra time allotted (intervention group 2) 4. Standard care for CST at the youth clinic with extra time allotted and the RLP-information (intervention group 3)

Step 2-4 will be conducted during different time periods at the same youth clinics. Recruitment for each step will be ongoing until the necessary number of participants are reached. All participating providers will be carefully instructed during educational sessions and provided with material on how to inform their visitors about the study. The providers at youth clinics will also receive oral information regarding how to execute the intervention and written materials (intervention guide, checklist) to ensure uniformity. During the project period, all providers will approach all adolescents visiting for CST and keep log over the visits to enable analysis of non-participants.

Participating adolescents in all groups will be asked to complete digital questionnaires after their visit. Primary outcomes: knowledge and awareness of CST, cervical cancer, fertility, and preconception health. Secondary outcomes: experience of the visit and likelihood to contact a midwife regarding questions about sexual or reproductive health in the future.

The power calculation is based on results by Stern et al. (2013) showing that university students increased knowledge by 40% after an RLP-intervention. The calculation assumed both greater variety in and lower increase in knowledge among adolescents than among university students. To detect a difference between the intervention and control group with 80% power and with a significance level of p< 0.05, 50 adolescents are needed in each group. We expect high participation rate and plan to recruit 75 adolescents in each group, i.e. 300 adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Persons with cervix
* 23 years of age
* Visiting midwife for their first cervical screening test

Exclusion Criteria:

* Non-Swedish-speaking

Ages: 23 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Experience of CST | Day 1. The patients receives a QR-code to the digital questionnaire at the end of the visit and can choose when and were to fill out the questionnaire, but are encouraged to do so in the waiting room
  The outcome is measured through self-reported data, collected through a digital questionnaire. The items are developed based on Kvalitet Ur Patientens Perspektiv (KUPP), which is a widely used measure within Swedish health care to measure PREM- Patient Reported Experience Measures

SECONDARY OUTCOMES:
Knowledge of and attitudes towards CST and cervical cancer | Day 1. The patients receives a QR-code to the digital questionnaire at the end of the visit and can choose when and were to fill out the questionnaire, but are encouraged to do so in the waiting room
  The outcome is measured through self-reported data, collected through a digital questionnaire. The item is developed based on previous research regarding knowledge of and attitudes towards CST and cervical cancer. The item is posed as 13 statements and the respondent is asked to tick the alternative that apply to her opinion: highly agree, partially agree, neither agree nor diagree, partially disagree, highly disagree, don't know.
Attitude towards contacting a midwife regarding sexual and reproductive health in the future | Day 1. The patients receives a QR-code to the digital questionnaire at the end of the visit and can choose when and were to fill out the questionnaire, but are encouraged to do so in the waiting room
  The outcome is measured through self-reported data, collected through a digital questionnaire. The item is formulated as the following "If you have questions about sexual and reproductive health in the future, how likely are you to turn to…midwife at the youth clinic? midwife at the midwifery clinic? nurse/doctor at the health center? 1177/UMO/YOUMO?" With the response alternatives: Very likely / Fairly likely / Neither likely nor unlikely / Fairly unlikely / Very unlikely
Knowledge of and attitudes towards fertility and preconception health | Day 1. The patients receives a QR-code to the digital questionnaire at the end of the visit and can choose when and were to fill out the questionnaire, but are encouraged to do so in the waiting room
  The outcome is measured through self-reported data, collected through a digital questionnaire. The item is developed based on the Health Belief Model and previous research on knowledge of and attitudes towards fertility and preconception health.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Stern, PhD, Principal Investigator — Uppsala University
Locations (1):
- Region Sörmland, Eskilstuna, Sweden

IPD SHARING:
Plan to Share IPD: No